CLINICAL TRIAL: NCT00457730
Title: A Randomized Placebo Controlled Trial of Duloxetine for Central Pain in Multiple Sclerosis
Brief Title: A Study to Test the Use of Duloxetine for Pain in MS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Theodore R Brown, Principle Investigator, Brown, Theodore R., M.D., MPH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1083575; WIRB Protocol Number: 20061712 (Other: Western IRB)
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Duloxetine; Pain
MeSH Terms: conditions — Multiple Sclerosis; Pain | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): subjects will be randomized to study drug (Duloxetine) or Placebo. Subjects will take 30 mg (10 capsules) titrate up to 60 mg( 40 capsules) and titrate back down to 30 mg.
  Interventions: Drug: Duloxetine
- placebo (Placebo Comparator): matched placebo medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Patients will be randomly assigned to Duloxetine 30mg/d for 1 week, 60mg/d for 5 weeks and 30mg/d for 1 week or placebo for 7 weeks under double-blind conditions.
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Placebo — Subjects are randomized to either Duloxetine or Placebo
  Other Names: Sugar Pill
  Arms: placebo

SUMMARY:
Many patients with Multiple Sclerosis experience pain that is caused by the effects of MS on the nervous system.

The purpose of this study is to see if an investigational drug (Duloxetine) will reduce pain in subjects with MS.

The US Food and Drug administration (FDA) has approved this drug for use with depression or pain from diabetes.However, it is considered investigational for this study because it has not been approved for patients with MS.

This study will recruit patients with MS who have central pain which is 4 or greater on a scale of 1-10. Patients must have experienced pain for 2 months or longer prior to begining the study.The study will last 10 weeks, patients will be randomized either Duloxetine or placebo and will be carefully monitored throughout the study. Patients will keep pain/sleep diaries during the study period and will be provided Ibuprofen for pain control.

DETAILED DESCRIPTION:
Between 350,000 and 400,000 Americans have Multiple Sclerosis, a chronic neurological disease characterized by demyelination and axonal degeneration. Pain is an important symptom of MS, reported in 44% to 80% of patients.

Duloxetine is FDA apprBetween 350,000 and 400,000 Americans have Multiple Sclerosis, a chronic neurological disease characterized by demyelination and axonal degeneration. Pain is an important symptom of MS, reported in 44% to 80% of patients.

Duloxetine is FDA approved for use in treatment of diabetic painful neuropathy and depression. Since the analgesic mechanism of action of Duloxetine is believed to occur in the Central Nervous System, there is reason to believe that it may also be effective in central pain conditions, such as MS.

Our study design includes a 1:1 randomization of Duloxetine to placebo. We hypothesize that the Duloxetine group will experience reductions in the weekly 24 hour average and worst pain scores that exceed 1.5 and that are significantly greater than reductions achieved in the placebo group. We also hypothesize that Duloxetine will be well tolerated with no significant group differences in adverse effects, sleep and quality of life as measured by the SF-36 approved for use in treatment of diabetic painful neuropathy and depression. Since the analgesic mechanism of action of Duloxetine is believed to occur in the Central Nervous System, there is reason to believe that it may also be effective in central pain conditions, such as MS.

Our study design includes a 1:1 randomization of Duloxetine to placebo. We hypothesize that the Duloxetine group will experience reductions in the weekly 24 hour average and worst pain scores that exceed 1.5 and that are significantly greater than reductions achieved in the placebo group. We also hypothesize that Duloxetine will be well tolerated with no significant group differences in adverse effects, sleep and quality of life as measured by the SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS made at least 3 months prior based on McDonald or Proser criteria.
* Age over 17.
* Clinical stability defined as no MS exacerbation or change in disease modifying therapy for 90 days prior to screening.
* Daily pain attributed to MS, present for a minimum of 2 months prior to screening.
* Minimum baseline score of 4 on the 24-h Worst Pain Score rated on an 11 point (0-10) point Likert Scale within the identified region of central pain.

Exclusion Criteria:

* Pain that could not clearly be differentiated from causes other than Multiple Sclerosis, such as diabetic neuropathy, PVD, arthritis or other musculoskeletal condition, chronic headache, visceral pain.
* Transient pains such as dysesthetic L'Hermittes sign alone.
* Current or historical diagnosis of mania, bipolar disorder or psychosis.
* Concomitant use of monoamine oxidase inhibitors (MAOI) or thioridazine.(MAOI drug must be discontinued 14 days prior to enrollment. At least 5 days must have passed after study drug discontinuation before MAOI drug may be started.)
* Concomitant use of a serotonin reuptake inhibitor or venlafaxine or duloxetine within 4 weeks of baseline.
* Use of any analgesic medication except ibuprofen for neurogenic pain 7 days prior to the baseline visit and until study termination.
* Use of an opioid, marijuana or dronabinol within 7 days of baseline.
* Narrow angle glaucoma.
* Depression with suicidality.
* Substantial alcohol use. Because it is possible that Duloxetine and alcohol interact to cause liver injury, duloxetine should not be prescribed to patients with substantial alcohol use. Potential subjects will be asked how much alcohol they drink. If the answer is over 2 drinks a day this will generally constitute an exclusion.
* History of chronic hepatic insufficiency or ALT or AST> twice the upper limit of normal. Because it is possible thast Duloxetine may aggravate pre exisitng liver disease, duloxetine should not be prescribed to patients with chronic liver disease.
* Renal insufficiency (Creatinine Clearance , 30mL/minor serum creatinine > 1.9). Duloxetine is not recommended for patients with end stage renal disease (requiring dialysis) or severe renal impairment. Population PK analyses suggest that mild to moderate degrees of renal dysfunction (estimated CrCl 30-80ml/min)have no significant effect on Duloxetine clearance. We will calculate creatinine clearance using the Cockcroft-Gault calculation. This is the most common calculation used in FDA producy labeling: Males=(140-age)(wt in kg)(serum creatinine)(72). Females= malesx 0.85.
* Uncontrolled hypertention (SBP>180, DBP>105)
* Females who are breast feeding, pregnant, or have potential to become pregnant during the course of the study.(fertile and unwilling/unable to use effective contraceptive measures)
* Any other serious and/or unstable medical condition.
* Allergy to ibuprofen or any other non steroidal anti inflammatory drug (NSAID)
* Any history of peptic ulcer disease within 2 years or lifetime history of NSAID-associated gastritis or other toxicity.
* Patients taking low dose aspirin will be instructed to contact their primary physicianto ask whether they may safely discontinue aspirin while participating in this study. If the recommendation is to continue aspirin or if use of aspirin is for secondary prevention of arteriosclerotic disease, then they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD.MPH, Principal Investigator — Evergreen Healthcare
Locations (1):
- Evergreen Healthcare, Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: subjects will be randomized to study drug (Duloxetine) or Placebo. Subjects will take 30 mg (10 capsules) titrate up to 60 mg( 40 capsules) and titrate back down to 30 mg.
  Placebo: Patients will be randomly assigned to Duloxetine 30mg/d for 1 week, 60mg/d for 5 weeks and 30mg/d for 1 week or placebo for 7 weeks under double-blind conditions.
  Placebo: Subjects are randomized to either Duloxetine or Placebo
- Placebo: subjects will be randomized to study drug (Duloxetine) or Placebo. Subjects will take 30 mg (10 capsules) titrate up to 60 mg( 40 capsules) and titrate back down to 30 mg.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 18 | 20
Completed | 14 | 19
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: subjects will be randomized to study drug (Duloxetine) or Placebo. Subjects will take 30 mg (10 capsules) titrate up to 60 mg( 40 capsules) and titrate back down to 30 mg.
  Placebo: Patients will be randomly assigned to Duloxetine 30mg/d for 1 week, 60mg/d for 5 weeks and 30mg/d for 1 week or placebo for 7 weeks under double-blind conditions.
  Placebo: Subjects are randomized to either Duloxetine or Placebo
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.71 (9.97) | 56.33 (11.23) | 56.3 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Worst Pain Score
Description: Weekly mean of 24 hour Worst Pain Score, percent change from baseline. Range is 0-10 with 0= no pain and 10= worst possible pain.
Time Frame: at week 6
Measure: Mean (Standard Deviation); unit: percent reduction on 0-10 analog scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 14 | 18
percent reduction on 0-10 analog scale | -29.1 (20.4) | -11.5 (18.2)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

2. Secondary Outcome: Percent Change in Average Pain Score.
Description: Percent change in Weekly mean of 24 hour Average pain Score, Week 6 vs. baseline. Range is 0-10 with 0= no pain and 10= worst possible pain.
Time Frame: at week 6
Measure: Mean (Standard Deviation); unit: percent reduction on 0-10 analog scale
Groups:
- Duloxetine: ubjects will take 30 mg daily for 1 week, then 60 mg daily for 5 weeks, then titrate back down to 30 mg daily for 1 week.
- Placebo: matched placebo medication throughout 6 week observation period
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 14 | 18
percent reduction on 0-10 analog scale | -38.5 (29.1) | -10.4 (18.85)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

3. Secondary Outcome: Global Impression of Change
Description: global impression: "How do you feel about the effects of the medication over the past 7 days? 7 point scale, 7 = delighted, 1= terrible
Time Frame: Week 6 vs baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine: Patients will be randomly assigned to Duloxetine 30mg/d for 1 week, 60mg/d for 5 weeks and 30mg/d for 1 week
- Placebo: matched placebo medication with same periods
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 13 | 18
units on a scale | 4.77 (1.3) | 3.94 (1.16)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.074, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Duloxetine: Study drug, Duloxetine, 30 mg for 1 week, titrate up to 60 mg for 5 weeks and titrate back down to 30 mg for 1 week.
- Placebo: Placebo: Matching placebo drug for 7 weeks total
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 6/18 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=18) | Placebo (N=20)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — nausea
headache (Nervous system disorders) | 2 (2) | 2 (2) — headache
dizziness (Nervous system disorders) | 2 (2) | 0 (0) — dizziness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No